CLINICAL TRIAL: NCT02776319
Title: Effects of Non-invasive Brain Stimulation in Tobacco Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Shirley Fecteau, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015-465
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Tobacco Use Disorder
Keywords: Non-invasive brain stimulation; tobacco use disorder; craving
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Experimental): Non-invasive brain stimulation (active)
  Interventions: Device: Non-invasive brain stimulation (active)
- Sham/Placebo (Placebo Comparator): Non-invasive brain stimulation (sham)
  Interventions: Device: Non-invasive brain stimulation (sham)

INTERVENTIONS:
Device: Non-invasive brain stimulation (active) — Non-invasive brain stimulation (active)
  Arms: Active
Device: Non-invasive brain stimulation (sham) — Non-invasive brain stimulation (sham)
  Arms: Sham/Placebo

SUMMARY:
The objective of the study is to determine the effect of non-invasive brain stimulation on craving for tobacco and brain metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Tobacco use disorder (DSM-V)

Exclusion Criteria:

* Other psychiatric disorders
* Contraindication to non-invasive brain stimulation and MRI

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Tobacco craving | During experimentation
  Subjective craving scale

SECONDARY OUTCOMES:
Brain metabolites | During experimentation
  Magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Social, Québec, Quebec, Canada